CLINICAL TRIAL: NCT04126434
Title: Intervention of Air Pollution and Acute Coronary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, WeiHuang, Principal Investigator, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WeiHuang19
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Masks

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no masking (Sham Comparator): not wearing facemask
  Interventions: Device: mask
- masking (Active Comparator): wearing facemask
  Interventions: Device: mask

INTERVENTIONS:
Device: mask — facemask

SUMMARY:
To determine the effect of intervention of ambient air pollution on acute coronary syndrome patients.

DETAILED DESCRIPTION:
To investgate the effect of wearing facemasks to decreasing levels of exposure to ambient air on acute coronary syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoker of any type during past six months and living in a non-smoking household.
2. A diagnosis of myocardial infarction or unstable angina 7-90 days prior to signed informed consent.

Exclusion Criteria:

1. Unstable CV disorders including uncompensated heart failure, refractory angina, uncontrolled arrhythmias, critical valvular heart disease and severe hypertension.
2. A history of infection with human immunodeficiency virus.
3. History of malignancy including leukemia and lymphoma AND/OR any severe, life-threatening disease AND/OR history of drug abuse within the last 2 years.
4. Pregnancy or intent to get pregnant during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
vascular function | six months
  Systolic blood pressure and diastolic blood pressure measured by omron HBP-1300
autonomic nervous function | six months
  Twenty four-hour electrocardiograms and heart rate variability

CONTACTS AND LOCATIONS:
Overall Officials: Wei Huang, PhD, Principal Investigator — Peking University Health Science Center
Locations (1):
- Peking University ,School of Public Health, Beijing, Beijing Municipality, China